CLINICAL TRIAL: NCT01252069
Title: A Phase III, Multicentre, Clinical Study Investigating the Efficacy and Safety of Three Successive Periods of 3-month Open-label PGL4001 Treatment, Each Followed by Ten Days of Double-blind Treatment With Progestin or Placebo and a Drug-free Period Until Return of Menses, in Subjects With Myomas and Heavy Uterine Bleeding
Brief Title: PGL4001 Efficacy Assessment in Reduction of Symptoms Due to Uterine Leiomyomata (PEARLIII-extension Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGL09-027
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate; Progestins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): PGL4001 10mg (oral tablets) for 3 months followed by a period of 10 days of placebo (oral tablets) during 3 periods each ended by a drug free period until return of menses.
  Interventions: Drug: PGL4001, placebo, drug free period
- B (Experimental): PGL4001 10mg (oral tablets) for 3 months followed by a period of 10 days of progestin (oral tablets) during 3 periods each ended by a drug free period until return of menses.
  Interventions: Drug: PGL4001, progestin, drug free period

INTERVENTIONS:
Drug: PGL4001, placebo, drug free period — PGL4001 10mg once daily (oral tablets) for 3 months followed by a period of 10 days of placebo (oral tablets) during 3 periods each ending with a drug free period until return of menses.
  Other Names: Ulipristal acetate
  Arms: A
Drug: PGL4001, progestin, drug free period — PGL4001 10mg once daily (oral tablets) for 3 months followed by a period of 10 days of progestin Norethisterone acetate 10mg once daily (oral tablets) during 3 periods each ending with a drug free period until return of menses.
  Other Names: Ulipristal acetate
  Arms: B

SUMMARY:
This is the long-term extension of a phase III, efficacy and safety open-label (protocol PGL09-026) with PGL4001 10mg tablets once daily for three months, blinded towards the administration of progestin or placebo tablets after end of PGL4001 treatment.

This extension study consists of three periods of 3 months open-label PGL4001 treatment, each followed by ten days of double-blind treatment with progestin or placebo and then a period without treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed visit 6 of PGL09-026 study, 10 to 18 days after menstruation following end of treatment with PGL4001, and did not take medications forbidden by the protocol.

Exclusion Criteria:

* Subject has a large uterine polyp (> 2cm).
* Subject has one or more ovarian cysts ≥ 4cm diagnosed by ultrasound during PGL09-026 study.
* Subject has abnormal hepatic function at re-test.
* Subject has clinically significant abnormal findings at visit A or any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the subject's safety or interfere with study evaluations.
* Subject has a positive pregnancy test or is planning a pregnancy during the course of the study.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
percentage of subjects in amennorrhoea at the end of each PGL4001 treatment course received | From baseline to end of each PGL4001 treatment (3months treatment)

CONTACTS AND LOCATIONS:
Locations (18):
- Medical University Vienna, department of obstetrics and gynecology, Vienna, Austria
- Belgium (3):
  - Cliniques Universitaires Saint-Luc Gynécologie-Obstétrique, Brussels
  - CHR de la Citadelle Gynécologie-Obstétrique, Liège
  - Cliniques Universitaires UCL de Mont-Godinne Gynécologie-Obstétrique, Yvoir
- Poland (9):
  - Prywatna Klinika Polozniczo-Ginekologiczna, Bialystok
  - INVICTA Sp. Z o.o., Gdansk
  - Private practice, Katowice
  - Private practice, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie Klinika Ginekologii Onkologicznej i Ginekologii, Lublin
  - Private Practice, Warsaw
  - Private practice, Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Klinika Poloznictwa, Chorob Kobiecych i Ginekologii Onkologicznej, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocławiu, I Katedra i Klinika Ginekologii i Położnictwa, Wroclaw
- Spain (5):
  - Hospital Universitario Hebron, gynecology department, Barcelona
  - Clinica Ginecologica CEOGA, departamento de Ginecologia, Lugo
  - Private Practice, Madrid
  - HOSPITAL Universitario 12 de Octubre y Fundación de Investigación Biomédica Hospital 12 de Octubre Departamento de Ginecología, Madrid
  - CHIP (Complejo Hospitalario Integral Privado), Málaga

REFERENCES:
- [Derived] Donnez J, Vazquez F, Tomaszewski J, Nouri K, Bouchard P, Fauser BC, Barlow DH, Palacios S, Donnez O, Bestel E, Osterloh I, Loumaye E; PEARL III and PEARL III Extension Study Group. Long-term treatment of uterine fibroids with ulipristal acetate ☆. Fertil Steril. 2014 Jun;101(6):1565-73.e1-18. doi: 10.1016/j.fertnstert.2014.02.008. Epub 2014 Mar 12. PMID 24630081